CLINICAL TRIAL: NCT07254663
Title: Influence of Swallow Gel and Semi-solid Consistency on Medication Dysphagia: A Multicenter Observational Study
Brief Title: GEL & MEDication Dysphagia
Acronym: GELMED
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-2989
Record Dates: First submitted 2025-09-15; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Neurological Diseases or Conditions; Healthy Participants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- neurogenic dysphagia group: patients with neurological diseases that may lead to dysphagia
  Interventions: Other: medication swallowing

INTERVENTIONS:
Other: medication swallowing — Three swallow trials will be conducted in randomized order for each of the following conditions:
  1. Placebo medication with methylene-blue-dyed water.
  2. Placebo medication with a semi-solid vehicle.
  3. Placebo medication with the swallowing gel GLOUP®.

SUMMARY:
This research project examines the prevalence of medication-related dysphagia in patients with dysphagia-associated diseases. Its primary aim is to assess how frequently swallowing difficulties occur during medication intake and to evaluate the impact of different consistencies-such as semi-solid formulations and commercial swallowing gels-on the swallowing process. Flexible endoscopic evaluation of swallowing serves as the diagnostic gold standard to determine whether alternative administration forms can facilitate safer swallowing. The findings are intended to support the optimization of medication intake and the prevention of complications in patients with dysphagia.

DETAILED DESCRIPTION:
Dysphagia refers to an impairment of the swallowing process, encompassing the transport of the food bolus from the oral cavity to the gastrointestinal tract. In neurological patients, combined disturbances of the oral and pharyngeal phases frequently occur, known as oropharyngeal dysphagia. This form of dysphagia not only significantly reduces quality of life but may also lead to severe complications.

A particularly relevant aspect of dysphagia is impaired swallowing of medication, referred to as medication dysphagia. This may compromise swallowing efficiency, for example when tablets or capsules remain in the oral cavity or pharynx and dissolve prematurely. Swallowing safety can also be affected, especially in cases of penetration or aspiration during medication intake.

To compensate for these difficulties, patients are often advised to swallow medication together with semi-solid substances instead of liquids. In addition, a commercially available swallowing gel has recently become accessible, designed specifically to facilitate medication intake in patients with dysphagia.

Despite its clinical relevance, medication dysphagia has rarely been investigated systematically with instrumental diagnostics. In particular, the compensatory strategies widely applied in practice have not yet been scientifically evaluated.

Objectives

This research project aims to determine the prevalence of medication dysphagia in patients with dysphagia-associated diseases and to assess the effects of different consistencies on the swallowing process. Specifically, the study will address the following questions:

What is the prevalence of medication dysphagia across different underlying diseases?

Is there an association between medication dysphagia and dysphagia for food and liquids?

How does the addition of a semi-solid vehicle affect the efficiency of medication swallowing?

How does the addition of a semi-solid vehicle affect the safety of medication swallowing?

How does the addition of a semi-solid vehicle influence subjective swallowing difficulties and swallowing-related anxiety during medication intake?

How does the use of a swallowing gel affect the efficiency of medication swallowing?

How does the use of a swallowing gel affect the safety of medication swallowing?

How does the use of a swallowing gel influence subjective swallowing difficulties and swallowing-related anxiety during medication intake?

Study Protocol

This is a prospective, multicenter interventional study. Eligible participants include patients with diseases associated with dysphagia who are scheduled for a clinically indicated Flexible Endoscopic Evaluation of Swallowing (FEES). Healthy control subjects will also be recruited for comparison.

At the University Hospital Düsseldorf, patients with neurovascular, neurodegenerative, neuroinflammatory, or neuromuscular diseases will be included. Medication dysphagia will be assessed using FEES. Three experimental paradigms are planned:

Standard FEES with food and liquid:

In the following order: 10 cc green-colored jelly (semi-solid), 10 cc methylene-blue-dyed liquid, and a piece of white bread (~3 × 3 × 0.5 cm, solid).

Three swallows will be tested for each bolus.

FEES assessment of medication dysphagia:

Three swallow trials will be conducted in randomized order for each of the following conditions:

1. Placebo medication with methylene-blue-dyed water.
2. Placebo medication with a semi-solid vehicle.
3. Placebo medication with the swallowing gel GLOUP®.

Subjective evaluation:

Perceived swallowing difficulty and swallowing-related anxiety will be assessed for each condition using a numerical rating scale (1-10).

Analysis

Medication dysphagia will be evaluated using a previously published and validated FEES-based classification system developed by our research group. This tool enables systematic assessment of swallowing efficiency and safety during medication intake.

ELIGIBILITY:
Inclusion Criteria:

Patients:

Adults with a dysphagia-associated disease (neurovascular, neurodegenerative, neuroinflammatory, or neuromuscular disorders; in other centers also ENT-related diseases), for whom FEES is clinically indicated.

Capable of providing informed consent and cognitively able to follow the study protocol.

Healthy Controls Adults without any dysphagia-associated disease (no neurovascular, neurodegenerative, neuroinflammatory, or neuromuscular disorders; no ENT-related diseases with structural abnormalities of the oropharynx or esophagus).

Capable of providing informed consent and cognitively able to follow the study protocol.

Exclusion Criteria:

No additional exclusion criteria beyond those specified in the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and relatives of the participating clinics
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Medication dysphagia score according to Labeit et al 2022; DOI: 10.1038/s41531-022-00421-9 | on the day of enrollment. This is not a longitudinal study but a one-time examination; all assessments take place on the day of enrollment.
Medication dysphagia swallowing score according to FEES (Labeit et al 2022; doi: 10.1038/s41531-022-00421-9) | on the day of enrollment. This is not a longitudinal study but a one-time examination; all assessments take place on the day of enrollment.
  as published here: Labeit et al 2022; doi: 10.1038/s41531-022-00421-9

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - University Hospital Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - University Hospital Münster, Münster, North Rhine-Westphalia
  - Hospital Osnabrücl, Onsabrück

IPD SHARING:
Plan to Share IPD: Yes
demographic data, clinical description of the cohort and swallowing results
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: beginning of recruitment until end of study